CLINICAL TRIAL: NCT00687674
Title: Phase I/II Study of Sorafenib, Lenalidomide, and Dexamethasone in Relapsed/Refractory Multiple Myeloma
Brief Title: Sorafenib, Lenalidomide, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to study design (and toxicity), this trial closed to accrual prior to opening the phase II portion.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000597065; P30CA015083 (NIH); MC078A (Other: Mayo Clinic); 07-006234 (Other: Mayo Clinic IRB); NCI-2009-01284 (Registry Identifier: NCI-CTRP); RV-MM-PI-0142 (Other: Celgene Protocol); SR06-933 (Other: Bayer Protocol)
Record Dates: First submitted 2008-05-30; First posted 2008-06-02 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Sorafenib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib + Lenalidomide + Dexamethasone (Experimental)
  Interventions: Drug: dexamethasone; Drug: sorafenib tosylate; Drug: Lenalidomide

INTERVENTIONS:
Drug: dexamethasone — 20 mg orally Days 1, 8, 15, 22 of 28 day cycle
Drug: sorafenib tosylate — Phase I - dose escalating: 200mg once daily dose level -2, 200mg once daily dose level -1, 200mg once daily dose level 0, 200mg twice daily dose level 1, 200mg twice daily dose level 2, 400mg AM & 200mg PM daily dose level 2a, 400mg twice daily dose level 3 orally days 1-28 every 28 days until progression
Drug: Lenalidomide — Phase I - dose escalating: 5mg level -2, 10mg level -1, 15mg level 0, 15mg level 1, 25mg level 2, 25mg level 2a, 25mg level 3 orally days 1-21 every 28 days until progression

SUMMARY:
RATIONALE: Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Sorafenib and lenalidomide may also stop the growth of cancer cells by blocking blood flow to the cancer. Giving sorafenib together with lenalidomide and dexamethasone may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of sorafenib when given together with lenalidomide and dexamethasone and to see how well they work in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of sorafenib tosylate and lenalidomide in combination with dexamethasone in patients with relapsed or refractory multiple myeloma. (phase I)
* To describe the toxicity of this regimen in these patients. (phase I)
* To evaluate the confirmed response in patients treated with this regimen. (phase II)

Secondary

* To correlate clinical effects (adverse events and/or tumor response or activity) with pharmacologic parameters (pharmacokinetics or pharmacodynamics) and/or biologic results (correlative laboratory). (phase II)
* To assess overall survival and time to disease progression in patients treated with this regimen. (phase II)

OUTLINE: This is a phase I, dose-escalation study of sorafenib tosylate in combination with lenalidomide followed by a phase II study.

Patients receive oral sorafenib tosylate once to twice daily on days 1-28, oral lenalidomide once daily on days 1-21, and oral dexamethasone on days 1, 8, 15, and 22. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and bone marrow sample collection periodically during study for laboratory correlative studies. Bone marrow plasma samples (i.e., fresh marrow aspirates) are assessed for marrow angiogenesis (microvessel density) by IHC; angiogenic capability (tubular network formation) by in vitro angiogenesis assay; tumor cell proliferation by bromo-2-deoxyuridine uptake; tumor cell apoptosis by three-color flow cytometry (CD38, CD45 or CD138, and 7AAD); and expression of VEGF and soluble VEGF receptors on plasma cells by enzyme-linked immunosorbent assay. Bone marrow biopsies are assessed for various phosphoproteins by IHC; phosphorylation status of ERK1/2 by immunoblotting; and for pharmacodynamic markers (e.g., P70 S6K) by immunoblotting. Blood samples are assessed for surface markers of circulating endothelial cells (CD105, CD34, and CD146) by flow cytometry and for circulating endothelial cell progenitors by late colony formation in mononuclear cells. The endothelial lineage is confirmed by phenotyping of surface markers for endothelial cells.

After completion of study therapy, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for phase I and 44 for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Relapsed or refractory disease requiring treatment
* Measurable disease, as defined by at least 1 of the following:

  * Serum monoclonal protein ≥ 1.0 g
  * More than 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30% (i.e., evaluable disease)
* No known standard therapy that is potentially curative for the patient's disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,000/μL
* Platelet count ≥ 75,000/μL
* Hemoglobin ≥ 9 g/dL
* Direct bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (≤ 5 times ULN if the liver is involved)
* Creatinine ≤ 2.5 times ULN
* Patients with treated or untreated POEMS (Patient-Oriented Evidence That Matters) allowed, provided they satisfy the criteria for measurable disease
* No other prior malignancy within the past year except currently treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, or prostate cancer not requiring therapy
* No other active malignancy requiring treatment that would interfere with the assessments of response of the myeloma to protocol treatment
* INR < 1.5 OR PT/PTT ≤ 1.5 times ULN

  * Patients receiving anticoagulation treatment with an agent such as warfarin or heparin are allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception for 28 days prior, during, and for 28 days after discontinuation of lenalidomide
* Willing to provide research samples according to the test schedule
* No uncontrolled infection
* No NYHA classification III or IV heart disease
* No unstable angina (i.e., anginal symptoms at rest), new-onset angina (i.e., began within the past 3 months), or myocardial infarction within the past 6 months
* No uncontrolled hypertension, defined as systolic blood pressure > 150 mm Hg or diastolic pressure > 90 mm Hg, despite optimal medical management
* No thrombotic or embolic events within the past 6 months, including cerebrovascular accidents and transient ischemic attacks
* More than 4 weeks since prior pulmonary hemorrhage or other bleeding event > grade 2
* No serious nonhealing wound or ulcer
* More than 4 weeks since prior significant traumatic injury
* No known positivity for HIV infection or infectious hepatitis, type A, B, or C
* No known hypersensitivity to thalidomide or lenalidomide
* No prior development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Able to take aspirin (325 mg) daily as prophylactic anticoagulation

PRIOR CONCURRENT THERAPY:

* Recovered from prior chemotherapy, regardless of interval since last treatment
* Prior lenalidomide therapy allowed
* More than 4 weeks since prior experimental therapy
* More than 4 weeks since prior major surgery or open biopsy
* No concurrent enrollment in any other study involving a pharmacologic agent or investigative therapy (i.e., drug, biologic, immunotherapy approaches, gene therapy) whether for symptom control or therapeutic intent
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (i.e., phenytoin, carbamazepine, and phenobarbital), rifampin, or Hypericum perforatum (St. John wort)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen (13) participants were recruited at Mayo Clinic between August 2008 and March 2010.
Pre-assignment Details: This was a phase I/II trial. A total of 13 participants were accrued, all to the phase I portion. This trial was terminated due to study design and toxicity during the phase I; therefore, the phase II portion will never open. No results from the phase II portion are available.
Period: Overall Study
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Started | 13
Completed | 11
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 13
Prior Lenalidomide [Number; unit: participants]
  Yes | 2
  No | 11
Prior Transplant [Number; unit: participants]
  Yes | 12
  No | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Grade 3 and 4 Adverse Event (Phase I)
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
  Description of Grades:
  Grade 1: Mild Grade 2: Moderate Grade 3: Severe Grade 4: Life-threatening Grade 5: Death
Time Frame: up to 3 years
Population: One participant refused further treatment prior to being assessed for adverse events.
Measure: Number; unit: participants
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 12
participants | 11

2. Primary Outcome: Number of Participants Who Achieve a Confirmed Response (Partial Response [PR], Very Good PR [VGPR], Complete Response [CR], or Stringent CR [sCR]) (Phase II)
Description: Response that was confirmed on 2 consecutive evaluations during treatment
  * CR: Complete disappearance of M-protein from serum & urine on immunofixation, <5% plasma cells in bone marrow (BM)
  * sCR: CR plus normal FLC ratio & absence of clonal cells in BM
  * VGPR: >=90% reduction in serum M-component; Urine M-Component <100 mg per 24 hours; <=5% plasma cells in BM
  * PR: >= 50% reduction in serum M-Component and/or Urine M-Component >= 90% reduction or <200 mg per 24 hours; or >= 50% decrease in difference between involved and uninvolved FLC levels
Time Frame: Duration on Treatment (up to 3 years)
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (Phase II)
Description: Overall Survival (OS) was defined as the time from registration to death of any cause. Participants were followed for a maximum of 2 years from registration. The median OS with 95%CI was estimated using the Kaplan Meier method
Time Frame: From registration to death (up to 3 years)
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Disease Progression (Phase II)
Description: Time to disease progression (TTP) was defined as the time from registration to progression. The median TTP with 95%CI was estimated using the Kaplan Meier method.
  Progression was defined as any one or more of the following:
  An increase of 25% from lowest confirmed response in:
  * Serum M-component (absolute increase >= 0.5g/dl)
  * Urine M-component (absolute increase >= 200mg/24hour
  * Difference between involved and uninvolved Free Light Chain levels (absolute increase >= 10mg/dl
  * Bone marrow plasma cell percentage (absolute increase of >=10%)
Time Frame: From registration to progression (up to 3 years)
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Microvessel Density From Baseline to Post-treatment and Correlation With > Clinical Outcomes (Phase II)
Time Frame: Pre and Post treatment (up to 3 years)
Reporting Status: Not Posted

6. Secondary Outcome: Change in Apoptosis Rate From Baseline to Post-treatment and Correlation With > Clinical Outcomes (Phase II)
Time Frame: Pre and Post treatment (up to 3 years)
Reporting Status: Not Posted

7. Secondary Outcome: Plasma Cell Gene Expression Profiles and Correlation With > Clinical Outcomes
Time Frame: Post treatment
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Stained Circulating Endothelial Cells and Endothelial Progenitor Cells and Correlation With Clinical Outcomes (Phase II
Time Frame: Post treatment
Reporting Status: Not Posted

9. Secondary Outcome: Change in VEGF Expression Levels and Correlation With Clinical Outcomes (Phase II)
Time Frame: Post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Sorafenib + Lenalidomide + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Lenalidomide + Dexamethasone (N=13)
Pneumonia (Infections and infestations) | 1 (1)
Leukopenia (Investigations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib + Lenalidomide + Dexamethasone (N=13)
Anemia (Blood and lymphatic system disorders) | 11 (53)
Diarrhea (Gastrointestinal disorders) | 4 (9)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral cavity Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 9 (63)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (6)
Infection without neutropenia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (5)
Bilirubin (Investigations) | 1 (1)
Leukopenia (Investigations) | 10 (64)
Lymphocyte count decreased (Investigations) | 1 (5)
Neutrophil count decreased (Investigations) | 10 (62)
Platelet count decreased (Investigations) | 10 (74)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (7)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (8)
Hypertension (Vascular disorders) | 4 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes